CLINICAL TRIAL: NCT00552422
Title: Domperidone for Gastroparesis Associated With Solid Organ Transplantation
Brief Title: Domperidone for Gastroparesis in Solid Organ Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of perceived need for domperidone in this population
Sponsor: David J. Lederer, M.D. (Other)
Responsible Party: Sponsor-Investigator, David J. Lederer, M.D., Herbert Irving Assistant Professor of Medicine and Epidemiology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAC3728
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Results first posted 2015-07-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-06

CONDITIONS: Gastroparesis; Gastroesophageal Reflux
Keywords: gastroparesis; gastroesophageal reflux
MeSH Terms: conditions — Gastroparesis; Gastroesophageal Reflux | interventions — Domperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Domperidone Arm (Experimental): Study subjects will self-administer oral domperidone 10mg four times a day. If symptoms persist for more than 7 days, the investigator may increase the dose to 20mg four times a day. 20mg four times a day will be the maximal dose. Subjects with signiﬁcant renal impairment will received a starting dose of 10mg twice a day. The maximal dose in subjects with signiﬁcant renal impairment will be 20mg twice a day.
  Interventions: Drug: domperidone

INTERVENTIONS:
Drug: domperidone — 10mg orally four times per day

SUMMARY:
The purpose of this study is to examine the clinical response to domperidone in solid organ transplant recipients with gastroparesis.

DETAILED DESCRIPTION:
After heart or lung transplantation, the stomach tends to empty much slower than normal. This slow emptying is called "gastroparesis." Gastroparesis is uncomfortable and often leads to nausea and vomiting. In addition to drastically impacting quality of life, severe nausea and vomiting can also lead to malnutrition and an inability to take oral medications, contributing to complications of transplantation. Treatments for gastroparesis include both medical and surgical therapies that work for some but not all patients.

Domperidone is a peripheral D2 antagonist that improves the emptying of the stomach in patients with gastroparesis. Domperidone is not FDA approved at this time. Some patients have developed lifethreatening abnormal heart rhythms after receiving domperidone intravenously. This problem has not been seen with domperidone given by mouth.

We propose to administer domperidone by mouth at standard doses to solid organ transplant patients who have gastroparesis that is not responsive to standard medical therapies or who experience adverse drug side effects. This study will not be blinded (open-label) and has a single treatment arm (no control or placebo group).

ELIGIBILITY:
Inclusion Criteria:

* gastroparesis or gastroesophageal reflux that is refractory to standard therapy.
* signed informed consent

Exclusion Criteria:

* serious cardiac arrhythmias
* clinically significant bradycardia, sinus node dysfunction, or heart block.
* prolonged QTc
* clinically significant electrolyte disorders.
* gastrointestinal hemorrhage or obstruction.
* prolactinoma
* pregnant or breast feeding female
* known allergy to domperidone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Lederer, M.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Domperidone Arm
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Domperidone Arm
Number analyzed (Participants) | 6
Age, Customized [Number; unit: participants]
  18-65 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Symptomatic Improvement
Description: The primary endpoint of the study is the achievement of a symptom grade of less then or equal to 3.
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | Domperidone Arm
Number analyzed (Participants) | 6
participants | 6

ADVERSE EVENTS:
Description: Adverse events were assessed systemically with routine ECG.
Groups:
- Domperidone: Participants ranged from 18-65 years of age. Gender composition was 60$% female and 40% male.
Arm/Group | Domperidone
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Domperidone (N=6)
long QTc (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No